CLINICAL TRIAL: NCT03627780
Title: Genetic Polymorphism Associated With the Occurrence of Postoperative Vomiting and Vomiting (PONV) in Patients Undergoing Oncological Surgeries
Brief Title: Genetic Polymorphism and Post Operative Nausea and Vomiting (PONV)
Acronym: ponv
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: NP1127/2017
Record Dates: First submitted 2018-08-09; First posted 2018-08-13 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Genetic Predisposition to Disease; Postoperative Nausea; Polymorphism, Genetic
MeSH Terms: conditions — Genetic Predisposition to Disease; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PONV: Patients presenting with postoperative nausea and vomiting
  Interventions: Diagnostic Test: DNA extraction
- no PONV: Patients not presenting with postoperative nausea and vomiting
  Interventions: Diagnostic Test: DNA extraction

INTERVENTIONS:
Diagnostic Test: DNA extraction — DNA will be extracted from white cells

SUMMARY:
Nausea and vomiting affects 25-30% of individuals in the post-operative period and can reach more than 70-80% in high-risk patients. inherited factors may play a significant role in individual susceptibility and clinical research on hereditary factors involved in the pathogenesis of Postoperative nausea and vomiting (PONV) and chemotherapy nausea and vomiting (CINV) is relatively new. The aim of this study is to investigate whether inter-individual differences related to PONV are associated with genetic factors. 300 patients will be evaluated in postoperative oncological surgeries. The peripheral leukocyte DNA will be extracted by the Salting Out Procedure method and processed to genotyping for 48 SNPs from 15 candidate genes by real-time PCR by the Taqman method. The possible associations with demographic data and factors related to surgery will be analyzed by univariate and multivariate analysis.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether inter-individual differences related to PONV are associated with genetic factors. 300 patients will be evaluated in postoperative oncological surgeries. The peripheral leukocyte DNA will be extracted by the Salting Out Procedure method and processed to genotyping for 48 single nucleotide polymorphisms (SNPs) from 15 candidate genes by real-time PCR by the Taqman method. The possible associations with demographic data and factors related to surgery will be analyzed by univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* High and intermediate-risk patients for PONV (Apfel score 2, 3 and 4)

Exclusion Criteria:

* Low risk patients for PONV (Apfel score 0 and 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 Patients submitted to cancer surgery, classified as high- and intermediate-risk for PONV according to Apfel Score, 150 cases and 150 controls.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
PONV (Post operative nausea and vomiting) | 24 hours
  Incidence of early (6 hours) and late (24 h) nausea and vomiting

SECONDARY OUTCOMES:
Intensity of Acute Postoperative pain | 24 hours
  Intensity of Postoperative pain measures by numerical rate scale and descriptive scale will be assessed in the first 24 hours in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Sousa, phd, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (2):
- Brazil (2):
  - Cancer Institute of the State of Sao Paulo - ICESP, São Paulo, São Paulo
  - Cancer Institute of the State of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
The researchers make a plan to share informations via Red Cap

REFERENCES:
- [Result] Hayase T, Sugino S, Moriya H, Yamakage M. TACR1 gene polymorphism and sex differences in postoperative nausea and vomiting. Anaesthesia. 2015 Oct;70(10):1148-59. doi: 10.1111/anae.13082. Epub 2015 May 27. PMID 26012530
- [Result] Wesmiller SW, Bender CM, Sereika SM, Ahrendt G, Bonaventura M, Bovbjerg DH, Conley Y. Association between serotonin transport polymorphisms and postdischarge nausea and vomiting in women following breast cancer surgery. Oncol Nurs Forum. 2014 Mar 1;41(2):195-202. doi: 10.1188/14.ONF.195-202. PMID 24578078
- [Derived] Grigio TR, Furuya TK, Slullitel A, Murillo Carrasco AG, Uno M, Alves MJF, Carmona MJC, Sugino S, Chammas R, Sousa AM. Clinical, ethnic and genetic risk factors associated with postoperative nausea and vomiting in patients undergoing cancer surgery: a case-control study. Am J Transl Res. 2025 Apr 15;17(4):3235-3246. doi: 10.62347/DGRM3907. eCollection 2025. PMID 40385041